CLINICAL TRIAL: NCT02649348
Title: Effects of Pre-operative Prehabilitation on the Clinical Outcomes of Gastric Cancer Patients With Metabolic Syndrome Who Undergo Laparoscopic Radical Gastrectomies: A Polit Randomized Clinical Trial
Brief Title: Effects of Prehabilitation in Gastric Cancer Patients With Metabolic Syndrome on Perioperative Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Yanbing Zhou, Professor, Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 81270449
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Stomach Neoplasms; Metabolic Syndrome X
Keywords: gastric neoplasm; metabolic syndrome; prehabilitation; pre-operative exercise; laparoscopic radical gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Metabolic Syndrome | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pre-operative prehabilitation (Other): Patients in the pre-operative prehabilitation group required the exercise intervention protocol, which included climbing six flights of stairs at least 6 times as a daily routine and adaptive simulated training of restrictive ventilation dysfunction following abdominal surgery by using a full elastic breathable abdominal bandage.
  Interventions: Behavioral: pre-operative prehabilitation
- Comparator (No Intervention): Patients in the control group did not need to undergo this pre-rehabilitation protocol and prepared conventionally.

INTERVENTIONS:
Behavioral: pre-operative prehabilitation — To climb six flights of stairs (approximately 20 meters in height) at least 6 times as a daily routine and adaptive simulated training of restrictive ventilation dysfunction (increased thoracic and decreased abdominal breathing compliance) following abdominal surgery by using a full elastic breathable abdominal bandage.
  Arms: pre-operative prehabilitation

SUMMARY:
A prospective randomised controlled trial to investigate the effects of a pre-operative prehabilitation protocol on clinical outcomes of gastric cancer patients with metabolic syndrome who undergo laparoscopic radical gastrectomies and to determine the underlying mechanisms.

DETAILED DESCRIPTION:
To investigate the effects of a pre-operative prehabilitation protocol on clinical outcomes of gastric cancer patients with metabolic syndrome who undergo laparoscopic radical gastrectomies and to determine the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* histologically-proven pre-operative stage I-III gastric cancer
* Combined with metabolic syndrome
* Age limits from 18 to 80 years old
* Classified into American Society of Anesthesiology (ASA) II or III surgical risk
* no history of abdominal surgery on organs located at the abdominal supramesocolic level

Exclusion Criteria:

* Combined with severe cardiac or pulmonary disease or other organ dysfunction
* ASA IV
* The history of abdominal surgery
* Conversion to open surgery
* The presence of gastrointestinal obstruction, perforation or necrosis;
* Declined to participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The proportion of postoperative complications | up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Han, M.D., Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No